CLINICAL TRIAL: NCT05893355
Title: The Effect of Acupressure Applied in the Late Postpartum Period After Cesarean Section on Back Pain
Brief Title: Non-Pharmacological Method to Relieve Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, sena dilek, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek4
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: Back Pain; Late postpartum; Cesarean Section
MeSH Terms: conditions — Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): * Participants in this group will be interviewed for the first time in the first week of postpartum and for the second time in the fourth week of postpartum. The application will be explained and a voluntary consent form will be signed.
  * Participant Information Form will be filled in by the researcher by face-to-face interview.
  * The VAS that will be applied to the participant to evaluate the back pain just before the application will be filled in by the participant.
  * The VAS Evaluating Back Pain after the application will be filled in by the participant.
  * The participant will be informed that the study has been completed.
  Interventions: Behavioral: Acupressure group
- Control group (No Intervention): * Participants in this group will be interviewed for the first time in the first week of postpartum and for the second time in the fourth week of postpartum. The application will be explained and a voluntary consent form will be signed.
  * Participant Information Form will be filled in by the researcher by face-to-face interview.
  * VAS to assess back pain will be filled in by the participant.
  * No application will be made to this group.

INTERVENTIONS:
Behavioral: Acupressure group — Application to Acupressure Group
  * Participants in this group will be interviewed for the first time at postpartum week 1, and for the second time between 4-6 weeks postpartum. The application will be explained and a voluntary consent form will be signed.
  * Participant Information Form will be filled in by the researcher by face-to-face interview.
  * The VAS, which will be applied to the puerperant women for the first time in the first week of the postpartum week and for the second time between the 4th-6th weeks, will be filled by the participant just before the application to evaluate the back pain.
  * The VAS Evaluating Back Pain after the application will be filled in by the participant.
  * The participant will be informed that the study has been completed.
  Arms: Acupressure group

SUMMARY:
The study will be carried out in a randomized controlled manner in order to examine the effectiveness of acupressure applied in the late postpartum period in postpartum women who have had back pain and have had a cesarean delivery. The sample of the study will consist of 70 participants who applied to the family health center between 05.06.2023 and 05.12.2024, who had cesarean birth registered in the central family health center in Kocaeli province Kandıra district, who met the research criteria and agreed to participate in the research. Data in the research; It will be collected using the 'Participant Information Form', 'VAS (Visual Analog Scale for Evaluating Back Pain)', 'McGill Pain Questionnaire (Short Form)'. Participants in the acupressure group will be given 2 times acupressure application in the 1st week and 4th week postpartum. No application will be made to the participants in the control group. The research is planned to be carried out after obtaining the necessary institutional and ethical committee permissions.

DETAILED DESCRIPTION:
Aim: The study was planned to examine the effect of acupressure on back pain in the late postpartum period after cesarean section.

Hypothesis(s):

H0: Acupressure application applied to puerperant women who had a cesarean delivery in the late postpartum period has no effect on reducing the level of back pain.

H1: Acupressure application applied to puerperant women who had cesarean delivery in the late postpartum period reduces the level of back pain.

Type of Research: This study was designed as a randomized controlled experimental study.

Research Population: The population of the research will consist of participants who have had cesarean section, who have back pain, who are in the late postpartum 1st week and 4th week, and who are registered to family medicine units in a Family Health Center.

It was calculated according to the research conducted by Akgün and Boz to determine the sample size in the study. The sample size of the study was calculated using the G*Power 3.1.9.2 program and the mean, standard deviation values and effect size of the back pain variable in the related article (Akgün & Boz, 2020) were taken into account. The effect size was calculated as 1.025136 by using the mean and standard deviation values of the related article. The minimum number of individuals to be included in the sample of the study to be done was calculated by taking G*Power 3.1.9.2 and effect size: 1.025136, α= 0.05, power: 0.90, and the sample size was determined as 23 in the acupressure group and 23 in the control group. A total of 70 (Acupressure group: 35, control group: 35 participants) participants will be included in the study, taking into account possible data losses.

In which group the participants included in the study will be, will be determined from the website of the random number generation program "Research Randomizer", and they will be divided into two groups. Thus, each participants's number and group number will be determined and recorded.

Data will be collected with the Introductory Information Form and VAS for assessing back pain.

Introductory Information Form: The form consists of a total of 31 questions questioning women's sociodemographic, obstetric, pregnancy-birth and postpartum back pain information. It is applied to the puerperant women for the first time in the postpartum 1st week and the second time in the postpartum 4th week.

VAS for Evaluation of Back Pain: The participant marks his or her own pain on a 10 cm ruler, which is marked as "no pain" at one end and the most severe pain at the other end. The participant is told that there are two endpoints and to mark any place between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

After obtaining the necessary ethics committee and institutional permissions for the implementation of the study, participants who had a cesarean section and who met the inclusion criteria of the study will be interviewed by going to the institution. Participants will be informed that they can participate in the study without affecting the care received at the family health center and they can leave the study at any time, and their voluntary consent will be obtained. After the participants are included in the study, they will be assigned to the study groups according to the electronic randomization table. The data will be collected by the researcher through face-to-face interviews at the family health center. VAS (Visual Analog Scale) will be filled in by the participants to evaluate late postpartum back pain. VAS (Visual analog scale) in which back pain is evaluated will be filled in the acupressure group and control group for the first time in the postpartum 1st week and the second time in the 4th week before and after the application. No application will be made to the control group and only routine care will be given.

An environment where privacy can be protected and away from external stimuli will be prepared for the participants. The application will be started by choosing the most comfortable position for the participants, leaving the application points open. For this study, 6 points (a total of 12 points on both sides from each point) were determined for this study, and these points are LI4, which is the 4th point of the large intestine meridian, Zhong Zu HT2 point, which is on the triple heater meridian, and Quchi, the 11th point of the large intestine meridian. /LI11, the 36th point of the stomach meridian is ST36, the 21st point of the gallbladder meridian is Jian Jing GB21, the 43rd point of the bladder meridian is UB 43. In addition, expert opinion was taken to determine the points. The practitioner will apply 15 seconds of warming, relaxing, and preparatory quality to the area of each of the notes, respectively, and lightly rubbing to reduce tension and tissue sensitivity. A total of 3 minutes will be spent preparing for all points. After the preparation, acupressure will be applied to each point for a total of 12 minutes for all points for 1 minute. Thumb, index and/or middle finger will be used in acupressure application. Consecutive, breathing rhythm compressions will be repeated without raising the finger. Repeated compressions will be at a frequency that does not disturb the person, does not cause pain and has a calming effect. Although there is a difference in the order of use of the determined acupressure points, this study will be carried out symmetrically to the LI4, HT2, LI11, ST36, GB21, UB43 points, respectively. The practitioner will have a stopwatch to control the time.

The data of the study will be evaluated using the Statistical Package for the Social Sciences (SPSS) 22.0 program. All data will first be evaluated with the Kolmogorov-Smirnov test for conformity to normal distribution, and then analyzed according to conformity to normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those suitable for normal distribution, median and minimum-maximum values for those that do not fit. Comparisons between groups for numerical variables of socio-demographic and clinical characteristics will be made with an independent two-sample t-test for normally distributed variables, and Mann-Whitney U test for non-normally distributed variables. Pearson Correlation test will be applied to determine the relationship between the fatigue severity of the experimental group and the tests and to determine the relationship between the tests. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years old,
* Able to read and write Turkish
* Postpartum 1st week and within 4th week
* Primiparous and multiparous
* Those who had a registered cesarean section in the family health center where the study was conducted,
* Able to speak and understand Turkish,
* Back pain score above 4 according to VAS (Visual analog scale),
* Participants who voluntarily agree to participate in the study will be included in the study.

Exclusion Criteria:

* Congenital anomaly in the baby who gave a stillbirth, whose baby is hospitalized in the neonatal intensive care unit,
* Use of cigarettes or alcohol
* History of past or present mental illness,
* Using antidepressants or anxiolytic drugs,
* With rheumatoid arthritis, ankylosing spondylitis, Scheuermann's disease, Ehlers-Danlos syndrome, spinal surgeries, nerve root compression, spondylolisthesis comorbid disease,
* Perineal edema, hematoma, wound dehiscence, bladder catheterization and serious postpartum complications (internal bleeding, femoral artery embolism, pelvic fracture),
* With impaired tissue integrity in the area to be applied,
* Vaginal delivery,
* Taking painkillers in the last 6 hours,
* In addition, those who want to leave the research at any stage of the research will be excluded from the research.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for assessing back pain | This scale will be filled by the participants before the application is made at the end of the first week after birth.
  The application will be made at the end of the first week after birth. The participant marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The participant is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.
Visual analog scale for assessing back pain | This scale will be filled in by the participants after the application is made at the end of the first week after birth.
  The application will be made at the end of the first week after birth. The participant marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The participant is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

SECONDARY OUTCOMES:
Visual analog scale for assessing back pain | This scale will be filled by the participants before the application is made at the end of the first mounth after birth.
  The application will be made at the end of the first mount after birth.. The participant marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The participant is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.
Visual analog scale for assessing back pain | This scale will be filled in by the participants after the application at the end of the first mounth after birth.
  The application will be made at the end of the first mount after birth.. The participant marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The participant is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mukerrem Sisman, Midwife, Study Chair — Kocaeli Kandıra Family Health Center
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No